CLINICAL TRIAL: NCT01031784
Title: Radioactive Holmium Microspheres for the Treatment of Patients With Non-resectable Liver Metastases of Mixed Origin; a Single Center, Interventional, Non-randomized, Open Label, Safety Study.
Brief Title: Radioactive Holmium Microspheres for the Treatment of Liver Metastases
Acronym: HEPAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, B.A. Zonnenberg, Principal investigator; MD, PhD, UMC Utrecht
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-450
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Liver Metastasis; Liver Tumors
Keywords: liver metastasis; Liver tumors; microspheres; holmium; toxicity
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Holmium-166 microspheres, intra-arterial (Experimental): intra-arterial administration of holmium-166 microspheres in the liver
  Interventions: Device: holmium-166 poly lactic acid microspheres; Device: holmium 166 microspheres

INTERVENTIONS:
Device: holmium-166 poly lactic acid microspheres — Intra arterial administration of radioactive Holmium 166 microspheres; 600 mg with a specific activity ranging from 1260 MBq per kilo liver weight to 5040 MBq in the highest dose
Device: holmium 166 microspheres — intra arterial administration of holmium 166 microsphers in the hepatic artery

SUMMARY:
The HEPAR study is aimed at determining the safety of radioactive holmium containing microspheres for the treatment of tumors in the liver. These microspheres will be administered by infusion in the liver artery using a arterial catheter in the femoral artery.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria may enter the study:

1. Patients must have given written informed consent.
2. Female or male aged 18 years and over.
3. Confirmed histological diagnosis of metastatic malignancy with dominant liver metastases without standard therapeutic options for treatment including chemotherapy or surgery. Dominant liver metastases are defined (according to the Response Evaluation Criteria in Solid Tumors (RECIST) methodology, see Appendix IV) as the diameter of all metastases in the liver must be more than 200% of the sum of the diameters of all soft tissue lesions outside the liver.
4. Life expectancy of 12 weeks or longer.
5. World Health Organisation (WHO) Performance status 0-2 (see Appendix III).
6. One or more measurable lesions at least 10 mm in the longest diameter by spiral Computed Tomography (CT) scan (5 mm slice thickness) according to the RECIST criteria.
7. Negative pregnancy test for women of childbearing potential. -

Exclusion Criteria:

Patients meeting any of the following criteria cannot enter the study:

1. Brain metastases or spinal cord compression, unless irradiated at least 4 weeks prior to the date of the experimental treatment and stable without steroid treatment for at least 1 week.
2. Radiation therapy within the last 4 weeks before the start of study therapy.
3. The last dose of prior chemotherapy has been received less than 4 weeks prior the start of study therapy.
4. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy.
5. Any unresolved toxicity greater than National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE version 3.0, see Appendix II) grade 2 from previous anti-cancer therapy.
6. Serum bilirubin > 1.5 x Upper Limit of Normal (ULN).
7. Serum creatinine > 185 µmol/L.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) > 5 x ULN.
9. Leukocytes < 4.0 109/l and/or platelet count < 150 109/l.
10. Significant cardiac event (e.g. myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
11. Pregnancy or breast feeding (women of child-bearing potential).
12. Comorbidity with a grave prognosis (estimated survival <3 months) and/or worse then the basic disease for which the patients will be included in the study.
13. Patients with abnormalities of the bile ducts (such as stents) with a increased chance of infections of the bile ducts.
14. Patients suffering from diseases with a increased chance of liver toxicity, such as primary biliary cirrhosis or xeroderma pigmentosum.
15. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
16. Patients who are declared incompetent.
17. Previous enrolment in the present study or previous treatment with radio-embolisation.
18. Treated with an investigational agent within 42 days prior to starting study treatment.
19. Female patients who are not using an acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) OR are less than 1 year postmenopausal or surgically sterile during their participation in this study (from the time they sign the consent form) to prevent pregnancy.
20. Male patients who are not surgically sterile or do not use an acceptable method of contraception during their participation in this study (from the time they sign the consent form) to prevent pregnancy in a partner.
21. Evidence of portal hypertension, splenomegaly or ascites.
22. Body weight over 150 kg.
23. Active hepatitis (B and/or C).
24. Liver weight > 3 kg (determined by software using CT data).
25. Allergy for i.v. contrast used (Visipaque®).
26. MRI contra-indications: severe claustrophobia, metal shrapnel, implanted pacemaker and/or neurostimulators.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Toxicity of Ho-166 poly lactic microspheres using CTC vs 3 criteria | 12 weeks

SECONDARY OUTCOMES:
tumor response according to RECIST criteria | 12 weeks
  tumor size will be determined using CT scans and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Zonnenberg, MD, Ph.D, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Vente MA, Nijsen JF, de Wit TC, Seppenwoolde JH, Krijger GC, Seevinck PR, Huisman A, Zonnenberg BA, van den Ingh TS, van het Schip AD. Clinical effects of transcatheter hepatic arterial embolization with holmium-166 poly(L-lactic acid) microspheres in healthy pigs. Eur J Nucl Med Mol Imaging. 2008 Jul;35(7):1259-71. doi: 10.1007/s00259-008-0747-8. Epub 2008 Mar 11. PMID 18330569
- [Background] Bult W, Vente MA, Zonnenberg BA, Van Het Schip AD, Nijsen JF. Microsphere radioembolization of liver malignancies: current developments. Q J Nucl Med Mol Imaging. 2009 Jun;53(3):325-35. PMID 19521312
- [Derived] Wagemans MEHM, Braat AJAT, van Rooij R, Smits MLJ, Bruijnen RCG, Prince JF, Bol GM, de Jong HWAM, Lam MGEH. Lung Mean Dose Prediction in Transarterial Radioembolization (TARE): Superiority of [166Ho]-Scout Over [99mTc]MAA in a Prospective Cohort Study. Cardiovasc Intervent Radiol. 2024 Apr;47(4):443-450. doi: 10.1007/s00270-023-03656-y. Epub 2024 Feb 7. PMID 38326577
- [Derived] Elschot M, Nijsen JF, Lam MG, Smits ML, Prince JF, Viergever MA, van den Bosch MA, Zonnenberg BA, de Jong HW. ((9)(9)m)Tc-MAA overestimates the absorbed dose to the lungs in radioembolization: a quantitative evaluation in patients treated with (1)(6)(6)Ho-microspheres. Eur J Nucl Med Mol Imaging. 2014 Oct;41(10):1965-75. doi: 10.1007/s00259-014-2784-9. Epub 2014 May 13. PMID 24819055
- [Derived] Smits ML, Nijsen JF, van den Bosch MA, Lam MG, Vente MA, Mali WP, van Het Schip AD, Zonnenberg BA. Holmium-166 radioembolisation in patients with unresectable, chemorefractory liver metastases (HEPAR trial): a phase 1, dose-escalation study. Lancet Oncol. 2012 Oct;13(10):1025-34. doi: 10.1016/S1470-2045(12)70334-0. Epub 2012 Aug 22. PMID 22920685
- [Derived] Smits ML, Nijsen JF, van den Bosch MA, Lam MG, Vente MA, Huijbregts JE, van het Schip AD, Elschot M, Bult W, de Jong HW, Meulenhoff PC, Zonnenberg BA. Holmium-166 radioembolization for the treatment of patients with liver metastases: design of the phase I HEPAR trial. J Exp Clin Cancer Res. 2010 Jun 15;29(1):70. doi: 10.1186/1756-9966-29-70. PMID 20550679